CLINICAL TRIAL: NCT05491798
Title: A Big Data-based Cohort Study for Cataract Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Clinical Professor, Sun Yat-sen University
Other Study IDs: CCPMOH2021-China-1
Record Dates: First submitted 2021-08-07; First posted 2022-08-08 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Cataract; Retina Disorder
Keywords: Cataract; Postoperative prediction; Image enhancement; Retina disorder
MeSH Terms: conditions — Cataract; Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Week
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Cataract is an important cause of blindness and visual impairment worldwide. At present, the only effective treatment method is surgery. The visual function of most patients can be significantly improved after surgery, but there are still 5-20% of patients whose visual function cannot be improved after surgery. Previous studies have found that the surgical complications and postoperative visual function of cataract patients are closely related to the condition of the fundus, but the current fundus camera cannot perform clear fundus imaging of cataract patients, and the existing potential visual inspections, such as retinal visual inspection, are also inaccurate. Predict postoperative visual acuity. Therefore, there is an urgent need for a reliable postoperative effect prediction system for cataract patients to provide reference for both ophthalmologists and patients.

This study intends to collect patient medical record information and traditional/ultra-wide fundus photos and other multi-modal data. Firstly, this study will use artificial intelligence technology to enhance fundus photos of cataract patients to obtain clearer fundus photos. Then this study will use both medical record information and traditional/ultra-wide fundus photographs to predict postoperative vision and visual function of cataract patients.

ELIGIBILITY:
Inclusion Criteria:

* Candidates for cataract surgery (phacoemulsification and intraocular lens implantation) within a week.

Exclusion Criteria:

* Unwilling or unable to receive fundus photography

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All candidates for cataract surgery (phacoemulsification and intraocular lens implantation) within a week.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Change of best corrected visual acuity | Baseline and 1 week after surgery
  Change of best corrected visual acuity from baseline to 1 week after surgery
Accuracy for detection of retinal disorders | 1 week after surgery
  Accuracy for detection of retinal disorders using enhanced fundus images

CONTACTS AND LOCATIONS:
Overall Officials: Haotian Lin, M.D., Ph.D., Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Liu L, Hong J, Wu Y, Liu S, Wang K, Li M, Zhao L, Liu Z, Li L, Cui T, Tsui CK, Xu F, Hu W, Yun D, Chen X, Shang Y, Bi S, Wei X, Lai Y, Lin D, Fu Z, Deng Y, Cai K, Xie Y, Cao Z, Wang D, Zhang X, Dongye M, Lin H, Wu X. Digital ray: enhancing cataractous fundus images using style transfer generative adversarial networks to improve retinopathy detection. Br J Ophthalmol. 2024 Sep 20;108(10):1423-1429. doi: 10.1136/bjo-2024-325403. PMID 38839251